CLINICAL TRIAL: NCT03102489
Title: Double-blind, Randomized, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BP101 After Multiple Doses Administration in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of BP101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ivix LLX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP101-HV02
Record Dates: First submitted 2017-03-13; First posted 2017-04-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hypoactive Sexual Desire Disorder(HSDD)
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP101 (Experimental): Treatment with BP101
  Interventions: Drug: BP101
- Placebo (Placebo Comparator): Treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP101 — Nasal spray
  Arms: BP101
Drug: Placebo — Nasal spray
  Arms: Placebo

SUMMARY:
Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of BP101 in Healthy Volunteers.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled study of the safety, tolerability, pharmacokinetics and pharmacodynamics of BP101 after multiple doses administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged from 18 to 40, inclusive.
* Verified diagnosis "healthy": absence gastrointestinal, hepatic, renal, cardiovascular, endocrine, central nervous system, ear, nose, throat (ENT) and gynecological disorders (performed standard clinical, laboratory and instrumental assessments did not reveal any disorders).
* Body mass index (BMI) within range from 18.5 to 30 kg/m^2.
* Subject consent not to intake alcohol during the entire study period; negative alcohol breath test at screening and before start of Investigational Product administration.
* Negative pregnancy test result at screening and before start of Investigational Product administration.
* Consent to use adequate methods of contraception throughout the study.
* Normal regular menstrual cycle of 28 +/- 7 days duration for at least 6 months before study enrollment.
* Women with stable sexual partner.

Exclusion Criteria:

* Chronic cardiovascular, respiratory, neuroendocrine, genitourinary systems disorders, as well as gastrointestinal, hepatic, renal, blood, and ENT disorders (including acute and chronic rhinitis, sinusitis, and others).
* Gynecological disorders (polycystic ovary syndrome, mommas, endometriosis, inflammatory diseases and others).
* Positive cervical cytology Papanicolaou (PAP) test in medical anamnesis within 12 months before screening.
* Lab abnormalities (blood hematology and biochemistry and urinalysis) at screening.
* Electrocardiogram (ECG) abnormalities at screening, and before start of Investigational Product administration.
* Systolic blood pressure in a sitting position below 100 mm Hg or above 140 mm Hg; and/or diastolic pressure below 60 mm Hg or above 90 mm Hg at screening and before start of Investigational Product administration.
* Heart rate less than 60 beats/min or more than 90 beats/min at screening, and before start of Investigational Product administration.
* Signs of malignant neoplasms in medical history, during the examination at any time prior to start of Investigational Product administration.
* Psychiatric disorders (including any form of schizophrenia, epilepsy, bipolar affective disorder and others), intake of psychotropic agents.
* Chronic pain syndromes (including chronic pelvic pain syndrome).
* Acute infections within 4 weeks before screening.
* Regular intake of medications (including nonprescription drugs, vitamins, and Supplements) within 2 weeks before screening.
* Intake of more than 5 units of alcohol per week (1 unit of alcohol is equivalent to 0.5 liter of beer, 200 ml wine or 30 ml of spirit (pure alcohol)) or historical information about alcoholism, substance abuse, prescription drug abuse.
* Smoking more than 10 cigarettes a day.
* Pregnancy or breastfeeding, positive urine pregnancy at screening and before the start of Investigational Product administration.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female healthy volunteers
Enrollment: 18 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events | 6 weeks
  To evaluate frequency, seriousness, and severity of adverse events, including events of dose-limiting toxicity in healthy volunteers receiving different doses of BP101 compared to placebo after multiple administrations.

SECONDARY OUTCOMES:
BP101 maximum plasma concentration (Cmax) | Day 1
  To determine pharmacokinetic parameter of maximum plasma concentration (Cmax) after single administration of BP101 in healthy volunteers.
BP101 area under the concentration versus time curve (AUC) | Day 1
  To determine pharmacokinetic parameter area under the plasma concentration versus time curve (AUC) after single administration of BP101 in healthy volunteers.
BP101 time to maximum plasma concentration (Tmax) | Day 1
  To determine pharmacokinetic parameter time to maximum plasma concentration (Tmax) after single administration of BP101 in healthy volunteers.
BP101 half-life time (T1/2) | Day 1
  To determine pharmacokinetic parameter of plasma half-life time (T1/2) after single administration of BP101 in healthy volunteers.
Change from Baseline in Female Sexual Function Index score | 2 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Female Sexual Function Index (FSFI).
Change from Baseline in Female Sexual Function Index score | 6 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Female Sexual Function Index (FSFI).
Change from Baseline in Female Sexual Distress Scale-Revised score | 2 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Female Sexual Distress Scale-Revised (FSDS-R).
Change from Baseline in Female Sexual Distress Scale-Revised score | 6 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Female Sexual Distress Scale-Revised (FSDS-R).
Change from Baseline in Female Sexual Function questionnaire score | 2 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Female Sexual Function (FSF) questionnaire.
Change from Baseline in Female Sexual Function questionnaire score | 6 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Female Sexual Function (FSF) questionnaire.
Change from Baseline in Arizona Sexual Experience Scale score | 2 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Arizona Sexual Experience Scale (ASEX) questionnaire.
Change from Baseline in Arizona Sexual Experience Scale score | 6 weeks
  To evaluate impact of BP101 in comparison with placebo on sexual function in healthy volunteers using Arizona Sexual Experience Scale (ASEX) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daniil Nemenov, M.D., Study Director — Ivix LLX
Locations (1):
- Research center Eco-Safety LLC, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No